CLINICAL TRIAL: NCT00436488
Title: Study of the Association Between ICAM-1 Polymorphisms and Severe Obesity
Brief Title: Frequency of ICAM-1 Polymorphisms in Obese Subjects
Status: Completed | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Other Study IDs: 12C501
Record Dates: First submitted 2007-02-16; First posted 2007-02-19 (Estimated); Last update posted 2007-02-19 (Estimated); Status verified 2007-02

CONDITIONS: Obesity
Keywords: ICAM-1; Obesity; Gene variants
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
The genetic contribution to the development of obesity is now well recognized. However obesity is a polygenic disease and thus many genes are likely to be involved. This study aims to investigate the possible association between specific variants of the gene coding for the Intercellular Adhesion Molecule-1 (ICAM-1)and the development of severe obesity in an Italian population

DETAILED DESCRIPTION:
Severely obese subjects referred to our institution will be evaluated. For the aim of the study, a venous blood sample will be obtained from these subjects and from a group of normal weight volunteers. Genomic DNA will be extracted from the blood samples and analysed by standard molecular biology techniques.The allelic and genotype frequencies of the two ICAM-1 variants will be calculated in the obese and control groups. The statistical significance of possible differences will be determined

ELIGIBILITY:
Inclusion Criteria:

* Obesity

Exclusion Criteria:

* Associated inflammatory diseases

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200
Dates: Start 2005-01; Study Completion 2006-07

CONTACTS AND LOCATIONS:
Overall Officials: Anna Maria Di Blasio, MD, Principal Investigator — Istituto Auxologico Italiano